CLINICAL TRIAL: NCT07253766
Title: The Effectiveness of Kinesiologic Taping in Patients With Knee Rheumatoid Arthritis in Terms of Pain, Function, and Kinesiophobia: A Randomised Controlled Trial
Brief Title: The Effectiveness of Kinesiologic Taping in Patients With Knee Rheumatoid Arthritis
Acronym: Taping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Rumeli University (Other)
Responsible Party: Principal Investigator, Ozden Baskan, Assist.Prof, Istanbul Rumeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E53938333-050-45035; Istanbul Rumeli University (Other: Istanbul Rumeli University)
Record Dates: First submitted 2025-09-18; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis; Pain; Kinesiophobia
Keywords: rheumatoid arthritis; pain; kinesiophobia; kinesiologic taping
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiologic taping group (Experimental): Kinesiology tape will be applied to the knee joint.
  Interventions: Other: kinesiologic taping
- Sham taping (Sham Comparator): Non-therapeutic sham taping will be applied to the knee joint
  Interventions: Other: sham taping

INTERVENTIONS:
Other: kinesiologic taping — The taping will be applied to the knee joint for 4 weeks.
  Arms: kinesiologic taping group
Other: sham taping — The non-therapeutic taping will be applied to the knee joint for 4 weeks.
  Arms: Sham taping

SUMMARY:
The goal of this clinical trial is to learn if kinesiologic taping works to treat individuals with Rheumatoid Arthritis.

The main questions it aim to answer:

* Is kinesiologic taping applied to the knee joint an effective treatment for pain, mobility, and kinesiophobia in individuals diagnosed with rheumatoid arthritis?
* Which is more effective? Kinesiologic taping or non-therapeutic sham taping? Which is better for pain, functional capacity, kinesiophobia and disease activity? Researchers will compare kinesiologic taping and non-therapeutic sham taping . Patients will be randomly divided into groups. The first group of patients was treated with sham taping, and the application period was applied consecutively for 4 weeks, with a minimum interval of 3 days and a maximum interval of 5 days. Group 2 patients underwent kinesiological taping, with the application period ranging from 3 to 5 days per week for 4 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 45 to 60
* Patients diagnosed with acute or chronic rheumatoid arthritis;
* Patients whose rheumatic medication protocol has not changed in the last 3 months; -Patients who do not smoke, drink alcohol or use drugs;
* Patients who have no vision, hearing or speech problems;
* Patients who are not amputees;
* Patients who can walk independently.

Exclusion Criteria:

* individuals over the age of 61;
* individuals with neurological disorders, severe chronic obstructive pulmonary disease, liver or kidney failure, malignancies, uncontrolled diabetes mellitus, major psychiatric disorders, or pregnancy; and those with concomitant conditions that could cause balance problems.
* Pregnant and breastfeeding women;
* individuals who had undergone surgery in the last few months;
* patients with loss of cooperation (e.g., those diagnosed with dementia or Alzheimer's disease) were also excluded from the study.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Four Weeks
  A Visual Analog scale(VAS) was used to assess pain intensity. Participants were asked to rate their perceived pain on a 10-cm horizontal line, where 0 cm indicates "no pain" and 10 cm indicates "worst pain imaginable." The participants marked a point on the line that best represented their pain intensity at rest and during activity. The distance (in centimeters) from the "no pain" end to the participant's mark was measured and recorded as the VAS score.
Tampa Kinesiophobia Scale | Four Weeks
  Kinesiophobia was assessed using the Tampa Scale for Kinesiophobia (TSK), a self-report questionnaire designed to measure fear of movement or re-injury. The scale consists of 17 items, each rated on a 4-point Likert scale ranging from 1 ("strongly disagree") to 4 ("strongly agree"). Higher scores indicate a greater degree of kinesiophobia, with a total score range between 17 and 68 points.
Timed up and Go test | Four weeks
  Functional mobility was assessed using the Timed Up and Go (TUG) test, a simple and reliable measure of dynamic balance and mobility. Participants were instructed to rise from a standard chair, walk three meters, turn around, walk back, and sit down at their normal walking speed. The time taken to complete the task was measured in seconds using a stopwatch. Shorter completion times indicate better functional mobility.
Disease Activity | Four weeks
  Disease activity was evaluated using the Disease Activity Score-28 (DAS28), which incorporates the number of tender and swollen joints (out of 28), the erythrocyte sedimentation rate (ESR), and the patient's global health assessment (GH) on a 100-mm Visual Analog Scale. The DAS28 score was calculated according to the standard formula, with values below 2.6 indicating remission, 2.6-3.2 low disease activity, 3.2-5.1 moderate activity, and above 5.1 high disease activity. This index is widely used to monitor disease progression and treatment response in patients with rheumatoid arthritis.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Rumeli University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT07253766/Prot_SAP_000.pdf